CLINICAL TRIAL: NCT01497886
Title: Randomized Controlled Trial Effect of Novel Intervention to Improve Stroke Symptom Recognition
Brief Title: Effect of Intervention to Improve Stroke Recognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Olajide Williams, Associate Professor of Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAF3455; 1R01NS067443-01A1 (NIH)
Record Dates: First submitted 2011-12-16; First posted 2011-12-23 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: Stroke; Children; Hip Hop Stroke; New York City
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Hop Stroke educational program (Active Comparator): Hip Hop Stroke is a school-based educational program that incorporates educational hip hop music and two cartoons to communicate stroke knowledge to children.
  Interventions: Behavioral: Hip Hop Stroke educational program
- Nutrition Education program (Placebo Comparator): The investigators will use what they will refer to as a "usual care" control. For this purpose the investigators have selected nutrition, physical activity, and obesity education. A trained facilitator will conduct the control program in the school auditorium. The investigators will use this control method to control for "attention", i.e., having a facilitator come to the classroom for the same amount of time as in the intervention that is, 1-hour sessions on three consecutive days. The facilitator will provide focused lectures on relevant topics, and show two short, 4-minute animated films on nutrition, and physical activity. The investigator will conduct parallel pretests and post-tests on the children (same as intervention testing sequence).
  Interventions: Behavioral: Nutrition Education program

INTERVENTIONS:
Behavioral: Hip Hop Stroke educational program — Three one-hour sessions, conducted over three consecutive days
  Arms: Hip Hop Stroke educational program
Behavioral: Nutrition Education program — The investigators will use what they will refer to as a "usual care" control. For this purpose the investigators have selected nutrition, physical activity, and obesity education. A trained facilitator will conduct the control program in the school auditorium. The investigators will use this control method to control for "attention", i.e., having a facilitator come to the classroom for the same amount of time as in the intervention that is, 1-hour sessions on three consecutive days. The facilitator will provide focused lectures on relevant topics, and show two short, 4-minute animated films on nutrition, and physical activity. The investigator will conduct parallel pretests and post-tests on the children (same as intervention testing sequence).
  Arms: Nutrition Education program

SUMMARY:
Despite the abundance of stroke education materials available, studies continue to reveal severe deficiencies in stroke literacy (knowledge of symptoms, urgent action, and prevention measures). Expensive mass media stroke education campaigns are not sustainable for this purpose, particularly in economically disadvantaged populations. Instead, the investigators propose to intervene in school classrooms with children aged 9 to 11 years, to teach the five cardinal stroke symptoms, the correct course of action when they occur, and to highlight the potential therapeutic benefit of early hospital arrival, with the intent that the children will then educate their parents. To help accomplish this, the investigators have developed a program called Hip Hop Stroke (HHS), which is comprised of rap songs and two animated musical cartoons that incorporate stroke knowledge.

DETAILED DESCRIPTION:
Stroke is the leading cause of serious long-term adult disability in the U.S. and third leading cause of death, and has a 2-fold greater incidence in Blacks compared to the majority Americans. Thrombolytic revascularization treatment administered within a maximum of 3 hours from symptom onset reduces morbidity, mortality and cost; however, only 3% of patients arrive at the hospital within 3 hours,4 mostly due to the public's lack of knowledge concerning stroke symptoms, and the appropriate response when they are recognized, which is to call 911. The investigators propose to reduce these delays using a novel behavioral intervention to improve symptom recognition and response in a high-risk, minority, economically disadvantaged population. Despite the abundance of stroke education materials available, studies continue to reveal severe deficiencies in stroke literacy (knowledge of symptoms, urgent action, and prevention measures). Expensive mass media stroke education campaigns are not sustainable for this purpose, particularly in economically disadvantaged populations. Instead, the investigators propose to intervene in school classrooms with children aged 9 to 11 years, to teach the five cardinal stroke symptoms, the correct course of action when they occur, and to highlight the potential therapeutic benefit of early hospital arrival, with the intent that the children will then educate their parents. To help accomplish this, the investigators have developed a program called Hip Hop Stroke (HHS), which is comprised of rap songs and two animated musical cartoons that incorporate stroke knowledge.

Targeting children to intervene with their parents has been rarely and sporadically attempted in various content areas, but the interventions have used traditional teaching methods that do not engage the children, and little success has been reported. In contrast, the HHS intervention was designed in collaboration with school-aged children, children's education television/media experts, as well as public health experts, school principals, and neurologists. As a result, not only is the targeting of children for this purpose an important innovation, but so is the careful development of materials designed to appeal to them. Moreover, the investigators note that utilizing children as a "transmission vector" for carrying out interventions aimed at their parents has the potential to serve as the basis for intervention in any number of other areas, for example, medication adherence, healthy eating and weight loss, treatment of diabetes, and so on.Thus, the significance of the proposed trial addresses the public health problem under study stroke symptom identification and response as well as development and refinement of a more general model of intervention.

ELIGIBILITY:
Inclusion Criteria:

* 4th-6th grade children and their parents in selected elementary public schools in the same geographical region/community with similar socioeconomic status (SES) and Ethnic composition.

Exclusion Criteria:

* School located in Harlem, New York.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4614 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2015-06-23 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Stroke Symptom and Response Knowledge Assessment (student) | Up to 3 days from baseline
  Knowledge of stroke prevention measures will be assessed by 8 YES/NO questions: 5 real and 3 distracters: eating lots of fruits and vegetables, exercising everyday, always taking medications given by doctor for high blood pressure/diabetes/high cholesterol, smoking avoidance or cessation, avoiding drug abuse, exercising once-a-week, eating lots of red meat, adding salt to meals.
Assessment of child's communication to parent regarding stroke symptoms. | Up to 7 days from baseline
  This measure assesses whether the child has talked with one of the adults in the household about what the child learned in school in both the HHS and control arms concerning symptoms of stroke and correct response.

SECONDARY OUTCOMES:
Assessment of events, latency to arrival at the emergency room. | 12 months from completion, and every 12 months afterwards
  The investigators will ask the participating parents to report any diagnosis of stroke received, at 12 months, continuing through the duration of the funding period. If the parent reports a stroke,the investigators will ask for permission to conduct a chart review to confirm the stroke diagnosis, and the treatment given (especially regarding thrombolytic therapy. The investigators will also ask the patient (or family member if the patient is non verbal), who recognized the symptoms (self or other or child) and who called 911.
Longitudinal Stroke Symptom and Response Knowledge Assessment (student) | 3 months after participation
  Knowledge of stroke prevention measures will be assessed by 8 YES/NO questions: 5 real and 3 distracters: eating lots of fruits and vegetables, exercising everyday, always taking medications given by doctor for high blood pressure/diabetes/high cholesterol, smoking avoidance or cessation, avoiding drug abuse, exercising once-a-week, eating lots of red meat, adding salt to meals.

CONTACTS AND LOCATIONS:
Overall Officials: Olajide A. Williams, MD MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams O, DeSorbo A, Noble J, Shaffer M, Gerin W. Long-term learning of stroke knowledge among children in a high-risk community. Neurology. 2012 Aug 21;79(8):802-6. doi: 10.1212/WNL.0b013e3182661f08. Epub 2012 Aug 8. PMID 22875089
- [Background] Williams O, DeSorbo A, Noble J, Gerin W. Child-Mediated Stroke Communication: findings from Hip Hop Stroke. Stroke. 2012 Jan;43(1):163-9. doi: 10.1161/STROKEAHA.111.621029. Epub 2011 Oct 27. PMID 22033995
- [Derived] Williams O, Leighton-Herrmann Quinn E, Teresi J, Eimicke JP, Kong J, Ogedegbe G, Noble J. Improving Community Stroke Preparedness in the HHS (Hip-Hop Stroke) Randomized Clinical Trial. Stroke. 2018 Apr;49(4):972-979. doi: 10.1161/STROKEAHA.117.019861. PMID 29567762